CLINICAL TRIAL: NCT06447571
Title: The Effect of Trunk Rehabilitation Compared to Core Stability on Balance, Gait, Falls and Community Mobility in Patients With Multiple Sclerosis
Brief Title: Trunk Rehabilitation Compared to Core Stability in Patients With Multiple Sclerosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Shatha Mukhtar, Principle Investigator, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Trunk Rehabilitation in MS
Record Dates: First submitted 2024-04-17; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Multiple Sclerosis; Trunk; Physical Therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Core Stability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: First visit, a blinded physiotherapist will evaluate the patient, then they will be randomly divided into two groups using a computer-generated system.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trunk Group (Experimental): Trunk exercises in multiplanar movement coupled with dual tasks on unstable surfaces.
  Interventions: Other: Trunk Rehabilitation
- Core stability Group (Active Comparator): Standard Core stability exercises carried in one plane on stable surfaces without dual tasks.
  Interventions: Other: Core Stability

INTERVENTIONS:
Other: Trunk Rehabilitation — Activating and strengthening the trunk muscles.
  Arms: Trunk Group
Other: Core Stability — Standard core stability fucus on lower trunk.
  Arms: Core stability Group

SUMMARY:
BACKGROUND Balance, gait, community mobility, and risk of falls are often associated with trunk impairment among people with Multiple Sclerosis (PwMS). Consequently, there is a pressing need for interventions addressing these concerns and exploring the potential effects of trunk rehabilitation.

LONG-TERM GOAL Offering guidance for effective plan selection, potentially included in rehabilitation guidelines for PwMS.

HYPOTHESIS Trunk exercises performed in multiplanar movement on unstable surfaces incorporated with dual-tasks (DT) could improve the functional outcomes more than standard one-plane core stability exercises.

SPECIFIC AIMS Investigating the effectiveness of trunk rehabilitation in PwMS and determining the optimal intervention strategy.

METHODS 50 PwMS randomly assigned into two groups. Trunk Group received trunk exercises on unstable surfaces with DT training, while the Core Group underwent standard one-plane core stability exercises on stable surfaces without DT. Additionally, both received conventional treatment. Primary outcome was the trunk impairment scale (TIS). Secondary outcomes included the Berg balance scale (BBS), Timed Up and Go (TUG), Modified Falls Efficacy (FES), Modified Fatigue Impact Scale (MFIS), Hospital Anxiety and Depression Scale (HADS), and Reintegration to Normal Living Index (RNLI).

SIGNIFICANCE Enhancing our understanding of trunk exercises' benefits and providing valuable guidance to clinicians for choosing the optimal treatment plan.

DETAILED DESCRIPTION:
There is a lack of comprehensive trunk rehabilitation protocols within the field of multiple sclerosis. The existing studies mostly focus on core stability, pelvic muscles, or alternative methods. Consequently, the aim was to develop a protocol to investigate the potential positive effects of trunk rehabilitation. Drawing from our review of relevant literature, investigators in this study have developed a trunk training protocol that focuses on multiplanar movements carried out on unstable surfaces and additionally, incorporated dual-task training (DT), which adds a layer of complexity.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with MS (McDonald's criteria)
* Able to walk 5 meters without assistance.
* No relapse in the past 2 months.

Exclusion Criteria:

* Recent surgery.
* Cognitive or psychological dysfunctions.
* Diagnosis of any other systematic disease.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Trunk Impairment Scale (TIS) | Baseline, 6 weeks, 1 month follow up.
  evaluates motor impairment of the trunk by assessing static and dynamic sitting balance and coordination of trunk movement. The total scores range between 0 for a minimal performance to 23 for a maximum performance.

SECONDARY OUTCOMES:
Berg Balance Scale (BBS) | Baseline, 6 weeks, 1 month follow up.
  standardized assessment tool utilized to objectively evaluate an individual's ability to maintain balance during specific tasks. The total scores range between 0 for a minimal performance to 56 for a maximum performance.
Timed Up and Go (TUG) | Baseline, 6 weeks, 1 month follow up.
  used to evaluate functional mobility.
Modified Falls Efficacy Scale (MFES) | Baseline, 6 weeks, 1 month follow up.
  modified and expanded version of the Falls Efficacy Scale (FES), which assesses the fear of falling. The total scores range between 0 reflecting less confidence and more fear of falling to 140 for more confidence and less fear of falling.
Modified Fatigue Impact Scale (MFIS) | Baseline, 6 weeks, 1 month follow up.
  evaluates the effects of fatigue on cognitive, psychosocial, and physical functioning. The total scores range from 0 reflecting less impact of fatigue to 84 for greater impact of fatigue.
Reintegration to Normal Living Index (RNLI) | Baseline, 6 weeks, 1 month follow up.
  to assess community mobility. focus on measuring the extent of reintegration into regular social activities among individuals affected by disease. Scores range from 0 to 110, a lower score indicates minimal integration, and higher scores indicate better integration. A total score out of 110 points is proportionally converted to create a score out of 100.

CONTACTS AND LOCATIONS:
Overall Officials: Majed M Albadi, PhD, Principal Investigator — King Abdulaziz University
Locations (1):
- King Abdulaziz University, Jeddah, Saudi Arabia

REFERENCES:
- [Derived] Mukhtar S, Aljohani G, Bakkar M, Almutairi N, Mazi A, Alsweed L, Albadi M, Aldhabi R, Khan F. The effects of trunk rehabilitation on balance, gait, falls, and community mobility in patients with multiple sclerosis: A single-blind randomized controlled trial. Mult Scler Relat Disord. 2025 Dec 13;106:106929. doi: 10.1016/j.msard.2025.106929. Online ahead of print. PMID 41421012